CLINICAL TRIAL: NCT00666978
Title: Enhancing Tobacco Use Treatment for African American Light Smokers
Brief Title: Health Education Counseling With or Without Bupropion in Helping African Americans Stop Smoking
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lisa Sanderson Cox, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Lisa Sanderson Cox, PhD, Research Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10332; R01CA091912 (NIH); KUMC-HSC-10332; KUMC-070313
Record Dates: First submitted 2008-04-24; First posted 2008-04-25 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Bladder Cancer; Cervical Cancer; Esophageal Cancer; Gastric Cancer; Head and Neck Cancer; Kidney Cancer; Leukemia; Liver Cancer; Lung Cancer; Pancreatic Cancer; Tobacco Use Disorder
Keywords: bladder cancer; cervical cancer; esophageal cancer; gastric cancer; renal cell carcinoma; adult primary liver cancer; non-small cell lung cancer; small cell lung cancer; pancreatic cancer; hypopharyngeal cancer; laryngeal cancer; lip and oral cavity cancer; nasopharyngeal cancer; oropharyngeal cancer; paranasal sinus and nasal cavity cancer; adult acute myeloid leukemia; tobacco use disorder
MeSH Terms: conditions — Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Leukemia; Liver Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Tobacco Use Disorder; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Leukemia, Myeloid, Acute | interventions — Bupropion; Gene Expression Profiling; Polymerase Chain Reaction; Counseling; Early Intervention, Educational; Psychiatric Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupropion Arm (Experimental): Subjects undergo smoking cessation intervention and take bupropion.
  Interventions: Behavioral: smoking cessation intervention; Drug: bupropion hydrochloride; Genetic: gene expression analysis; Genetic: polymerase chain reaction; Other: counseling intervention; Other: educational intervention; Procedure: psychosocial assessment and care
- Health Education Arm (Placebo Comparator): Subjects receive counseling intervention and take placebo.
  Interventions: Behavioral: smoking cessation intervention; Genetic: gene expression analysis; Genetic: polymerase chain reaction; Other: counseling intervention; Other: educational intervention; Procedure: psychosocial assessment and care

INTERVENTIONS:
Behavioral: smoking cessation intervention
Drug: bupropion hydrochloride
  Arms: Bupropion Arm
Genetic: gene expression analysis
Genetic: polymerase chain reaction
Other: counseling intervention
Other: educational intervention
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: A stop-smoking plan that includes health education counseling and bupropion may help African-American smokers stop smoking. It is not yet known whether health education counseling is more effective with or without bupropion in helping African Americans stop smoking.

PURPOSE: This clinical trial is studying health education counseling and bupropion to see how well they work compared with a placebo and health education counseling in helping African Americans smokers stop smoking.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of bupropion hydrochloride and health education counseling vs placebo and health education counseling for smoking cessation among African Americans who are light smokers.

Secondary

* To characterize CYP2A6 activity in African Americans who are light smokers by evaluating phenotype (3'hydroxycotinine/cotinine ratio [3HC/COT]) and CYP2A6 genotype.
* To evaluate the relationship between CYP2A6 activity and smoking cessation outcomes.
* To evaluate CYP2A6 genetic polymorphisms associated with nicotine and cotinine metabolism in African Americans who are light smokers.
* To measure baseline cotinine and metabolite levels to evaluate the nicotine metabolism phenotype of 3HC/COT.
* To evaluate the relationship between nicotine metabolism phenotype of 3HC/COT and smoking cessation outcomes.
* To evaluate CYP2A6 genotype as a predictor of smoking cessation outcomes.

Tertiary

* To characterize CYP2B6 activity in African Americans who are light smokers by evaluating phenotype and CYP2B6 genotype.
* To evaluate the relationship between CYP2B6 activity and smoking cessation outcomes.
* To measure steady state bupropion hydrochloride and metabolite levels to identify a bupropion metabolism phenotype.
* To evaluate the relationship between bupropion hydrochloride metabolism phenotype and smoking cessation outcomes.
* To evaluate the relationship between CYP2B6 genetic polymorphisms (genotype) and blood levels of bupropion hydrochloride and active metabolites (phenotype).
* To determine the effects of CYP2B6 genotype as predictors of smoking cessation outcomes.

OUTLINE: Participants are randomized to one of two arms.

* Arm I: Participants receive oral bupropion hydrochloride once or twice daily in weeks 0-6. Participants also undergo 6 sessions of health education counseling conducted in person during clinic visits in weeks 0, 3, and 7 and via telephone in weeks 1, 5, and 16. The health education counseling sessions include providing information about the risks of continued smoking and the benefits of quitting, developing a quit plan, outlining a concrete quit day preparation plan, discussing strategies for successful quitting, building social support, reducing stress, recognizing and managing withdrawal and craving, overcoming barriers to abstinence, and using medication for smoking cessation. Participants receive Kick It at Swope: Stop Smoking Guide, a culturally-sensitive smoking cessation guide, to review with their study counselor during the first counseling session.
* Arm II: Participants receive an oral placebo once or twice daily in weeks 0-6. Participants also undergo health education counseling as in arm I.

Participants complete baseline questionnaires about demographics, smoking history, and psychometrics, including the following: racial identity, depressive symptoms, alcohol use, stress, smoking consequences, social support, environmental influences of smoking, adherence to study medication, nicotine withdrawal, craving, and mood.

Participants undergo serum sample collection in weeks 0 and 3. To standardize the time since the last cigarette, participants are asked to smoke one cigarette prior to serum sample collection in week 0. Samples are analyzed for nicotine metabolism phenotype and bupropion hydrochloride metabolism phenotype by liquid chromatography and mass spectrometry and CYP2A6 and CYP2B6 genotype by polymerase chain reaction and polymorphism analysis. Participants who self-report abstinence also undergo saliva sample collection in weeks 7 and 26 to measure cotinine levels to verify smoking status.

After completion of study intervention, participants are followed at 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* African American who has smoked ≤ 10 cigarettes per day for ≥ 2 years AND has smoked for ≥ 25 days within the past month

  * Not a heavy smoker
  * No other forms of tobacco within the past 30 days
* Must be interested in stopping smoking
* No other smoker in the household enrolled in this study

PATIENT CHARACTERISTICS:

* Has a home address and a functioning telephone number
* Not planning to move from the Kansas City metro area within the next 12 months
* Not pregnant or nursing
* Negative pregnancy test
* No alcohol or substance abuse within the past year
* Not currently drinking ≥ 14 alcoholic drinks per week
* No binge drinking (5 or more drinks on one occasion) on at least two occasions within the past month
* No history of seizures or head trauma
* No history of bulimia or anorexia nervosa
* No myocardial infarction within the past 30 days
* No reported use of opiates, cocaine, or stimulants
* No diabetes requiring oral hypoglycemics or insulin

PRIOR CONCURRENT THERAPY:

* More than 30 days since prior nicotine replacement therapy, fluoxetine, clonidine, buspirone, or doxepin
* No other concurrent medication that contains bupropion hydrochloride
* No concurrent psychoactive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2007-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa S. Cox, PhD, Principal Investigator — University of Kansas
Locations (2):
- United States (2):
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Swope Health Central, Kansas City, Missouri

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Chenoweth MJ, Peng AR, Zhu AZX, Cox LS, Nollen NL, Ahluwalia JS, Benowitz NL, Knight J, Swardfager W, Tyndale RF. Does sex alter the relationship between CYP2B6 variation, hydroxybupropion concentration and bupropion-aided smoking cessation in African Americans? A moderated mediation analysis. Addiction. 2022 Jun;117(6):1715-1724. doi: 10.1111/add.15742. Epub 2021 Dec 3. PMID 34791718
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] El-Boraie A, Chenoweth MJ, Pouget JG, Benowitz NL, Fukunaga K, Mushiroda T, Kubo M, Nollen NL, Sanderson Cox L, Lerman C, Knight J, Tyndale RF. Transferability of Ancestry-Specific and Cross-Ancestry CYP2A6 Activity Genetic Risk Scores in African and European Populations. Clin Pharmacol Ther. 2021 Oct;110(4):975-985. doi: 10.1002/cpt.2135. Epub 2021 Jan 1. PMID 33300144
- [Derived] Nollen NL, Mayo MS, Ahluwalia JS, Tyndale RF, Benowitz NL, Faseru B, Buchanan TS, Cox LS. Factors associated with discontinuation of bupropion and counseling among African American light smokers in a randomized clinical trial. Ann Behav Med. 2013 Dec;46(3):336-48. doi: 10.1007/s12160-013-9510-x. PMID 23733379
- [Derived] Clausius RL, Krebill R, Mayo MS, Bronars C, Martin L, Ahluwalia JS, Cox LS. Evaluation of the brief questionnaire of smoking urges in Black light smokers. Nicotine Tob Res. 2012 Sep;14(9):1110-4. doi: 10.1093/ntr/ntr267. Epub 2012 Jan 12. PMID 22241828
- [Derived] Berg CJ, Cox LS, Choi WS, Mayo MS, Krebill R, Bronars CA, Ahluwalia JS. Assessment of depression among African American light smokers. J Health Psychol. 2012 Mar;17(2):197-206. doi: 10.1177/1359105311414953. Epub 2011 Jul 20. PMID 21775497
- [Derived] Cox LS, Faseru B, Mayo MS, Krebill R, Snow TS, Bronars CA, Nollen NL, Choi WS, Okuyemi KS, Salzman GA, Benowitz NL, Tyndale RF, Ahluwalia JS. Design, baseline characteristics, and retention of African American light smokers into a randomized trial involving biological data. Trials. 2011 Jan 25;12:22. doi: 10.1186/1745-6215-12-22. PMID 21266057

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupropion Arm: 270 African American adults received bupropion (150mg bid) for 7 weeks in addition to health education counseling.
- Placebo Arm: 270 African American adults received placebo for 7 weeks in addition to health education counseling.
Period: Overall Study
Arm/Group | Bupropion Arm | Placebo Arm
Started | 270 | 270
Completed | 192 | 187
Not Completed | 78 | 83

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion Arm | Placebo Arm | Total
Number analyzed (Participants) | 270 | 270 | 540
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (11.1) | 46.2 (11.5) | 46.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 183 | 357
  Male | 96 | 87 | 183
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 270 | 270 | 540
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 270 | 270 | 540
Married or living with partner [Count of Participants; unit: Participants] — Population: One participant refused the question.
  Participants
    number analyzed (Participants) | 269 | 270 | 539
    (all) | 91 | 75 | 166
Monthly family income <$1800 [Count of Participants; unit: Participants] — Population: 6 participants refused the question.
  Participants
    number analyzed (Participants) | 267 | 267 | 534
    (all) | 169 | 158 | 327
Education > or = high school [Count of Participants; unit: Participants] — Population: One participant refused the question.
  Participants
    number analyzed (Participants) | 269 | 270 | 539
    (all) | 225 | 229 | 454
Weight [Mean (Standard Deviation); unit: lbs] | 196.1 (51.8) | 194.8 (54.0) | 195.5 (52.9)
BMI [Mean (Standard Deviation); unit: kg/m 2] — Population: One participant refused to collect weight.
  kg/m 2
    number analyzed (Participants) | 269 | 270 | 539
    (all) | 31.1 (7.6) | 31.1 (8.1) | 31.1 (7.9)
Depression(CESD-10) score [Mean (Standard Deviation); unit: units on a scale] — CESD-10 assessed distress associated with depressive symptoms: possible total score ranges from 0 to 30, with a score of 10 or greater reflecting clinically significant depression. Population: One participant refused the questions.
  units on a scale
    number analyzed (Participants) | 269 | 270 | 539
    (all) | 7.2 (4.9) | 8.2 (5.5) | 7.7 (5.2)
Stress (PSS-4) [Mean (Standard Deviation); unit: units on a scale] — PSS-4 assessed self-appraised global stress: possible total score ranges from 0 to 16. Higher scores indicate more stress. Population: One participant refused to answer.
  units on a scale
    number analyzed (Participants) | 269 | 270 | 539
    (all) | 4.9 (3.1) | 5.5 (3.3) | 5.2 (3.2)
Serum Cotinine [Mean (Standard Deviation); unit: ng/ml] — Population: 4 participants had samples that were unable to be analyzed.
  ng/ml
    number analyzed (Participants) | 269 | 267 | 536
    (all) | 268.7 (160.2) | 283.0 (151.2) | 275.8 (155.8)
Exhaled Carbon monoxide [Mean (Standard Deviation); unit: ppm] — Population: Exhaled carbon monoxide was added after the study began and was collected only on 411 of 540 participants.
  ppm
    number analyzed (Participants) | 202 | 209 | 411
    (all) | 15.8 (9.4) | 17.1 (10.5) | 16.4 (10.0)
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 8.0 (2.6) | 7.9 (2.4) | 8.0 (2.5)
Fagerstrom Test for Nicotine Dependence- 6 item [Mean (Standard Deviation); unit: score] — FTND assessed nicotine dependence: possible total score ranges from 0 to 10. 0 indicates minimum physical nicotine dependence and 10 indicates maximum physical nicotine dependence.
  score | 3.1 (1.7) | 3.3 (1.7) | 3.2 (1.7)
Time to first cigarette,< or = 30 minutes [Count of Participants; unit: Participants] | 191 | 199 | 390
Smoke Menthol Cigarettes [Count of Participants; unit: Participants] | 224 | 228 | 452
Quit Attempts [Mean (Standard Deviation); unit: Quit Attempts] — Number of 24-hour quit attempts made in the past year.
  Quit Attempts | 3.5 (7.9) | 3.9 (7.4) | 3.7 (7.7)
Pharmacotherapy use during most recent quit attempt [Count of Participants; unit: Participants] | 72 | 61 | 133
Age of first cigarette [Mean (Standard Deviation); unit: years] | 17.5 (5.8) | 18.1 (7.3) | 17.6 (5.9)
Age started smoking regularly [Mean (Standard Deviation); unit: years] — Population: One participant declined to respond.
  years
    number analyzed (Participants) | 269 | 270 | 539
    (all) | 21.1 (6.7) | 21.3 (7.4) | 21.1 (7.1)
Motivation Scale [Mean (Standard Deviation); unit: units on a scale] — Motivation to quit smoking scale asking about how important it is to quit smoking in the next week. 1 item scale. Scale of 0 = not important and 10 = extremely important.
  units on a scale | 9.7 (0.8) | 9.8 (0.7) | 9.7 (0.8)
Confidence Scale [Mean (Standard Deviation); unit: units on a scale] — Confidence to quit smoking scale asking about how confident you are that you could quit smoking completely in the next week. 1 item scale. Scale of 0 = not confident and 10 = extremely confident.
  units on a scale | 7.9 (2.1) | 7.8 (2.0) | 7.9 (2.4)
Smoke-free household [Count of Participants; unit: Participants] | 65 | 67 | 132
California Tobacco Survey: Inhale deeply [Count of Participants; unit: Participants] — Question asks "Which statement best describes how or whether you inhale?" Response options include 'I inhale deeply into my chest', I inhale partly into my chest', I inhale as far back as my throat', 'I inhale back into my throat', 'I just puff, I don't really inhale'.
  Reporting number of participants who answered 'I inhale deeply into my chest'.
  Participants | 65 | 61 | 126

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Salivary Cotinine-verified Smoking Abstinence at 6 Months
Description: Salivary cotinine-verified smoking abstinence at 6 months. A cut point of 15 ng/ml was used to differentiate smokers from nonsmokers.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bupropion Arm | Placebo Arm
Number analyzed (Participants) | 270 | 270
Participants | 36 | 27
Statistical Analysis 1: Comparison: Bupropion Arm vs Placebo Arm; Based on our previous studies, sample size was determined a priori assuming a two-sided x2 test with a type I error rate of .05, a power of 80%, and a cotinine-verified abstinence rate of 15% in the placebo group and 25% in the bupropion SR group at week 26, with the assumption that those lost to follow-up would be imputed as smokers; Test type: Superiority — The x2 test was used to determine whether there was a difference between treatment groups (bupropion SR vs placebo) in verified 7-day point prevalence abstinence at week 26, imputing the missing participants as smokers; p = .23, t-test, 2 sided — All tests of statistical significance were two-sided, and all P values less than .05 were considered statistically significant; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.82 to 2.35] — Raw proportions were used to estimate the verified cessation rate in each group and corresponding odds ratio along with its 95% confidence interval

2. Secondary Outcome: Number of Slow and Fast Metabolizers by Metabolite Ratio
Description: Analyzed CYP2A6 by activity, called the nicotine metabolite ratio using a split between slow and fast metabolism at 0.31.
  The variants present in people in the slow genotype group include *17, *20, *23,*27, *35, *9, *2, *25, *26, and *4. The fast metabolizers have none of the variant alleles tested.
  Blood samples were collected for 3HC/COT ratio at Week 0.
Time Frame: Weeks 0
Population: This variant is related to nicotine metabolism and was collected from all study participants but not analyzed by study arm as it does not relate to the study medication. Data pre-specified to be collected and reported as a single arm.
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: All study participants were African American adults and received either bupropion (150mg bid) for 7 weeks in addition to health education counseling or placebo for 7 weeks in addition to health education counseling.
Arm/Group | All Study Participants
Number analyzed (Participants) | 450
Participants
  Fast Metabolizers by Nicotine Metabolite Ratio | 236
  Slow Metabolizers by Nicotine Metabolite Ratio | 214
Statistical Analysis 1: Comparison: All Study Participants; Test type: Other; p = 0.0022, Regression, Logistic — This reflects Week 7; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.95 to 0.99] — This reflects Week 7

3. Secondary Outcome: Number of Participants for Each CYP2B6 Allele
Description: We genotyped CYP2B6 in 268 from the Bupropion arm as this polymorphism is related to bupropion metabolism.
Time Frame: Week 3
Measure: Count of Participants; unit: Participants
Groups:
- Bupropion Arm: 270 African American adults received bupropion (150mg bid)for 7 weeks in addition to health education counseling.
Arm/Group | Bupropion Arm
Number analyzed (Participants) | 268
Participants
  CYP2B6*4 Allele Frequency | 2
  CYP2B6*5 Allele Frequency | 6
  CYP2B6*6 Allele Frequency | 95
  CYP2B6*9 Allele Frequency | 0
  CYP2B6*16 Allele Frequency | 0
  CYP2B6*18 Allele Frequency | 17
  CYP2B6*22 Allele Frequency | 6
Statistical Analysis 1: Comparison: Bupropion Arm; Test type: Other; p < 0.05, Regression, Linear — Analysis relied on examining quit rates using linear regression, where the hydroxybupropion was a significant predictor of smoking cessation. CYP2B6 genotype was not a direct significant predictor of cessation in either the placebo or bupropion arm; Odds Ratio (OR) = 2.82 — Bupropion adherent individuals with higher hydroxybupropion levels were more likely to be abstinent at Weeks 3, 7 and 26 compared to individuals with lower hydroxybupropion levels

4. Secondary Outcome: Number of Slow and Fast Metabolizers by Genotype
Description: Analyzed CYP2A6 by genotype. The variants present in people in the slow genotype group include *17, *20, *23,*27, *35, *9, *2, *25, *26, and *4. The fast metabolizers have none of the variant alleles tested.
  Slow metabolizers have any reduction or loss of function variant. Fast metabolizers are *1/*1 genotype by exclusion.
Time Frame: Week 0
Population: This variant is related to nicotine metabolism and was collected from all study participants but not analyzed by study arm as it does not relate to the study medication. Data pre-specified to be collected and reported as a single arm. Blood was unable to be analyzed for CYP2A6 genotype for 6 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 534
Participants
  Slow Metabolizers by Genotype | 265
  Fast Metabolizers by Genotype | 269

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Bupropion Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/270 | 0/270
Serious Adverse Events (participants affected / at risk) | 8/270 | 13/270
Other Adverse Events (participants affected / at risk) | 46/270 | 29/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion Arm (N=270) | Placebo Arm (N=270)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Infection, Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acoustic nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Coagulation (Cardiac disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 2 (2)
MIddle ear infection (Infections and infestations) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Personality Change (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion Arm (N=270) | Placebo Arm (N=270)
Headache (Nervous system disorders) | 9 (9) | 15 (15)
Insomnia (Psychiatric disorders) | 26 (26) | 9 (9)
Nausea (Gastrointestinal disorders) | 11 (11) | 5 (5)

LIMITATIONS AND CAVEATS:
Over half of the participants who expressed interest in this study were ineligible according to study protocol. The lack of assessment between standardized assessment points limited the ability to characterize the process of relapse.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes